CLINICAL TRIAL: NCT00847301
Title: Observational Cohort Study to Evaluate Safety and Efficacy of Pradaxa (Dabigatran Etexilate) in Patients With Moderate Renal Impairment (Creatinine Clearance 30-50 ml/Min) Undergoing Elective Total Hip Replacement Surgery or Total Knee Replacement Surgery
Brief Title: Pradaxa (Dabigatran Etexilate) 150 mg/q.d. in Patients With Moderate Renal Impairment After Hip or Knee Replacement Surgery
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.84
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-08

CONDITIONS: Arthroplasty, Replacement; Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Renal Impairment

SUMMARY:
An observational cohort study on safety and efficacy to generate additional data on the benefit/risk profile of the 150 mg dose of Pradaxa in patients with renal impairment

ELIGIBILITY:
Inclusion criteria:

Patients of 18 years of age or above with moderate renal impairment (creatinine clearance 30-50 ml/min) undergoing elective total hip replacement surgery who consent in writing to their participation in this observational study

Exclusion criteria:

All patients who should not be treated with Pradaxa 150 mg according to the European Summary of Product Characteristics (SPC):

severe renal impairment (creatinine clearance < 30 ml/min); elevated liver enzymes > 2 upper limit of normal (ULN); Hepatic impairment or liver disease expected to have any impact on survival, anaesthesia with post-operative indwelling epidural catheters, hypersensitivity to dabigatran etexilate or to any of the excipients, active clinically significant bleeding, organic lesion at risk of bleeding, spontaneous or pharmacological impairment of haemostasis, concomitant treatment with quinidine, protehetic heart valve requiring anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate renal insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2009-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (53):
- Austria (2):
  - 1160.84.4301 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.84.4310 Boehringer Ingelheim Investigational Site, Vienna
- France (20):
  - 1160.84.3311 Boehringer Ingelheim Investigational Site, Angers
  - 1160.84.3334 Boehringer Ingelheim Investigational Site, Bordeaux
  - 1160.84.3303 Boehringer Ingelheim Investigational Site, Caen
  - 1160.84.3314 Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 1160.84.3320 Boehringer Ingelheim Investigational Site, Créteil
  - 1160.84.3307 Boehringer Ingelheim Investigational Site, Dijon Cédex
  - 1160.84.3310 Boehringer Ingelheim Investigational Site, Illkirch-Graffenstaden
  - 1160.84.3335 Boehringer Ingelheim Investigational Site, Le Havre
  - 1160.84.3326 Boehringer Ingelheim Investigational Site, Les Lilas
  - 1160.84.3312 Boehringer Ingelheim Investigational Site, Lyon
  - 1160.84.3305 Boehringer Ingelheim Investigational Site, Marseille
  - 1160.84.3323 Boehringer Ingelheim Investigational Site, Nantes Cédex 2
  - 1160.84.3302 Boehringer Ingelheim Investigational Site, Paris
  - 1160.84.3306 Boehringer Ingelheim Investigational Site, Paris
  - 1160.84.3313 Boehringer Ingelheim Investigational Site, Pierre-Bénite
  - 1160.84.3324 Boehringer Ingelheim Investigational Site, Poitiers Cédex
  - 1160.84.3322 Boehringer Ingelheim Investigational Site, Saint Etienne Cédex 2
  - 1160.84.3319 Boehringer Ingelheim Investigational Site, Saint-Saulve
  - 1160.84.3316 Boehringer Ingelheim Investigational Site, Toulouse Cédex 9
  - 1160.84.3332 Boehringer Ingelheim Investigational Site, Vannes Cédex
- Germany (11):
  - 1160.84.04903 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.84.04947 Boehringer Ingelheim Investigational Site, Erlangen
  - 1160.84.4922 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 1160.84.04927 Boehringer Ingelheim Investigational Site, Hachenburg
  - 1160.84.04929 Boehringer Ingelheim Investigational Site, Koblenz
  - 1160.84.04902 Boehringer Ingelheim Investigational Site, Marburg
  - 1160.84.04946 Boehringer Ingelheim Investigational Site, München
  - 1160.84.04913 Boehringer Ingelheim Investigational Site, Olsberg
  - 1160.84.04914 Boehringer Ingelheim Investigational Site, Sylt
  - 1160.84.04938 Boehringer Ingelheim Investigational Site, Wismar
  - 1160.84.04948 Boehringer Ingelheim Investigational Site, Würzburg
- Italy (4):
  - 1160.84.03908 Boehringer Ingelheim Investigational Site, Latina
  - 1160.84.03902 Boehringer Ingelheim Investigational Site, Milan
  - 1160.84.03904 Boehringer Ingelheim Investigational Site, Monza
  - 1160.84.03909 Boehringer Ingelheim Investigational Site, Udine
- Spain (8):
  - 1160.84.3409 Boehringer Ingelheim Investigational Site, Badalona (Barcelona)
  - 1160.84.3410 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.84.3403 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.84.3405 Boehringer Ingelheim Investigational Site, Málaga
  - 1160.84.3404 Boehringer Ingelheim Investigational Site, Pamplona
  - 1160.84.3412 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón - Madrid
  - 1160.84.3401 Boehringer Ingelheim Investigational Site, Valencia
  - 1160.84.3402 Boehringer Ingelheim Investigational Site, Zaragoza
- Sweden (3):
  - 1160.84.4603 Boehringer Ingelheim Investigational Site, Kungälv
  - 1160.84.4601 Boehringer Ingelheim Investigational Site, Motala
  - 1160.84.4604 Boehringer Ingelheim Investigational Site, Sollefteå
- United Kingdom (5):
  - 1160.84.04405 Boehringer Ingelheim Investigational Site, Basildon
  - 1160.84.04408 Boehringer Ingelheim Investigational Site, Bedford
  - 1160.84.04403 Boehringer Ingelheim Investigational Site, Luton
  - 1160.84.04401 Boehringer Ingelheim Investigational Site, Wigan
  - 1160.84.04407 Boehringer Ingelheim Investigational Site, Yeovil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 472 patients entered into the study, 428 were treated with moderate renal impairment. Treated patients with moderate renal impairment are presented.
Groups:
- Overall Study Design: All Patients treated with dabigatran etexilate (Pradaxa), planned dose: 75 mg at the day of surgery, from the day after surgery to last treatment day 150 mg once daily
Period: Overall Study
Arm/Group | Overall Study Design
Started | 428
Completed | 374
Not Completed | 54
Not completed — Adverse Event | 35
Not completed — Switch to other anticoagulants | 16
Not completed — Lost to Follow-up | 1
Not completed — No prescription after hospital discharge | 1
Not completed — Other reason not defined above | 1

BASELINE CHARACTERISTICS:
Population: The Treated set with moderate renal impairment: this patient set included all patients with CrCl (Creatinine clearance) 30 - 50 mL/min who received at least one 1 of dabigatran etexilate.
Groups:
- All Patients: All Patients treated with dabigatran etexilate (Pradaxa), planned dose: 75 mg at the day of surgery, from the day after surgery to last treatment day 150 mg once daily.
Arm/Group | All Patients
Number analyzed (Participants) | 428
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 324
  Male | 104

OUTCOME MEASURES:

1. Secondary Outcome: Documented Symptomatic Proximal DVT, Documented Symptomatic Distal DVT, Documented Symptomatic Nonfatal Pulmonary Embolism and All-cause Mortality
Description: Percentage of participant with documented symptomatic proximal DVT (deep vein thrombosis), documented symptomatic distal DVT, documented symptomatic nonfatal pulmonary embolism and all-cause mortality
Time Frame: From first intake (day of surgery) until 24 hours after last intake (planned: knee replacement: Day 10 after surgery, hip replacement: Day 28-35 after surgery) of Pradaxa
Population: Treated set with moderate renal impairment: this patient set included all patients with CrCl 30 - 50 mL/min who received at least one 1 of dabigatran etexilate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 428
percentage of participants
  symptomatic distal DVT | 0.23 [0.01 to 1.29]
  symptomatic proximal DVT | 0.0 [0.00 to 0.86]
  symptomatic non-fatal PE | 0.23 [0.01 to 1.29]
  All-cause mortality | 0.23 [0.01 to 1.29]

2. Primary Outcome: Percentage of Patients With Major Bleeding Events (MBE)
Description: Major bleeding events were defined according to the modified McMaster criteria, and were classified by the investigator as Major bleeding event or Any bleeding event. The criteria for MBE's were: fatal; clinically overt associated with loss of haemoglobin >=20g/L in excess of what was expected; clinically overt leading to the transfusion of >=2 units packed cells or whole blood in excess of what was expected; symptomatic retroperitoneal, intracranial, intraocular or intraspinal; requiring treatment cessation; leading to re-operation
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 428
percentage of participants | 2.10 [0.97 to 3.95]

3. Primary Outcome: Percentage of Patients With Symptomatic Venous Thromboembolic Events (sVTE) and All Cause Mortality
Description: The co-primary efficacy variable sVTE was defined as the composite of documented symptomatic proximal and distal deep vein thrombosis (DVT) and documented symptomatic non-fatal pulmonary embolism (PE) and All Cause Mortality.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | All Patients
Number analyzed (Participants) | 428
percentage of Participants | 0.70 [0.14 to 2.03]

4. Secondary Outcome: Percentage of Patients With Major Extra-surgical Site Bleedings
Description: Percentage of Patients With Major Extra-surgical Site Bleedings
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | All Patients
Number analyzed (Participants) | 428
percentage of Participants | 1.87 [0.81 to 3.65]

5. Secondary Outcome: Volume of Wound Drainage (Post-operative)
Description: Volume of Wound Drainage after surgery
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | All Patients
Number analyzed (Participants) | 428
ml | 685.2 (404.1)

ADVERSE EVENTS:
Time Frame: From first drug intake up to 24 h after last drug intake; planned number of days after surgery: knee replacement: 10 days, hip replacement: 28-35 days
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 34/468
Other Adverse Events (participants affected / at risk) | 24/468
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=468)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3
Catheter site haemorrhage (General disorders) | 1
Inflammation (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Arthritis infective (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Hepatic enzyme increased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Petit mal epilepsy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 2
Circulatory collapse (Vascular disorders) | 1
Haematoma (Vascular disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Scar (Injury, poisoning and procedural complications) | 1
Suture related complication (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Wound secretion (Injury, poisoning and procedural complications) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=468)
Vomiting (Gastrointestinal disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.